CLINICAL TRIAL: NCT02340936
Title: National, Open-label, Multicentre Phase I-II Study of Combination R-ESHAP With Lenalidomide as Salvage Therapy for Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma Candidates to Stem-cell Transplantation
Brief Title: Clinical Trial to Determinate Dose, Security and Efficacy or Lenalidomide and Rituximab (LR)-ESHAP in Patients With Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Collaborators: Celgene Corporation (Industry); Dynamic Science S.L. (Industry); Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LR-ESHAP
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2018-02

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LR-ESHAP (lenalidomide 5 mg) (Experimental): Intervention: lenalidome 5mg combined with R-ESHAP (3 cycles of treatment every 21 days: lenalidomide 5 mg/day (day 1 to 14 except cycle 2 that will be administered from day 1 to 10), etoposide 40 mg/m2/day (day 1 to day 4), methylprednisolone 500 mg/day (day 1 to day 5), cisplatin 25 mg/m2/day (day 1 to day 4), cytarabine 2000 mg/m2 (day 5) and rituximab 375 mg/m2 (day 1 or 5)).
  Interventions: Drug: LR-ESHAP (lenalidomide 5 mg)
- LR-ESHAP (lenalidomide 10mg) (Experimental): Intervention: lenalidome 10mg combined with R-ESHAP( 3 cycles of treatment every 21 days: lenalidomide 10 mg/day (day 1 to 14 except cycle 2 that will be administered from day 1 to 10), etoposide 40 mg/m2/day (day 1 to day 4), methylprednisolone 500 mg/day (day 1 to day 5), cisplatin 25 mg/m2/day (day 1 to day 4), cytarabine 2000 mg/m2 (day 5) and rituximab 375 mg/m2 (day 1 or 5)).
  Interventions: Drug: LR-ESHAP (lenalidomide 10 mg)
- LR-ESHAP (lenalidomide 15mg) (Experimental): Intervention: lenalidome 15mg combined with R-ESHAP (3 cycles of treatment every 21 days: lenalidomide 15 mg/day (day 1 to 14 except cycle 2 that will be administered from day 1 to 10), etoposide 40 mg/m2/day (day 1 to day 4), methylprednisolone 500 mg/day (day 1 to day 5), cisplatin 25 mg/m2/day (day 1 to day 4), cytarabine 2000 mg/m2 (day 5) and rituximab 375 mg/m2 (day 1 or 5)).
  Interventions: Drug: LR-ESHAP (lenalidomide 15 mg)
- LR-ESHAP (lenalidomide 20mg) (Experimental): Intervention: lenalidome 20mg combined with R-ESHAP (3 cycles of treatment every 21 days: lenalidomide 20 mg/day (day 1 to 14 except cycle 2 that will be administered from day 1 to 10), etoposide 40 mg/m2/day (day 1 to day 4), methylprednisolone 500 mg/day (day 1 to day 5), cisplatin 25 mg/m2/day (day 1 to day 4), cytarabine 2000 mg/m2 (day 5) and rituximab 375 mg/m2 (day 1 or 5)).
  Interventions: Drug: LR-ESHAP (lenalidomide 20 mg)

INTERVENTIONS:
Drug: LR-ESHAP (lenalidomide 5 mg) — 3 cycles of lenalidomide 5mg, etoposide, methylprednisolone, cisplatin, cytarabine and rituximab every 3 weeks.
  Other Names: LR-ESHAP
  Arms: LR-ESHAP (lenalidomide 5 mg)
Drug: LR-ESHAP (lenalidomide 10 mg) — 3 cycles of lenalidomide 10mg, etoposide, methylprednisolone, cisplatin, cytarabine and rituximab every 3 weeks.
  Other Names: LR-ESHAP
  Arms: LR-ESHAP (lenalidomide 10mg)
Drug: LR-ESHAP (lenalidomide 15 mg) — 3 cycles of lenalidomide 15mg, etoposide, methylprednisolone, cisplatin, cytarabine and rituximab every 3 weeks.
  Other Names: LR-ESHAP
  Arms: LR-ESHAP (lenalidomide 15mg)
Drug: LR-ESHAP (lenalidomide 20 mg) — 3 cycles of lenalidomide 20mg, etoposide, methylprednisolone, cisplatin, cytarabine and rituximab every 3 weeks.
  Other Names: LR-ESHAP
  Arms: LR-ESHAP (lenalidomide 20mg)

SUMMARY:
The purpose of the Phase I of the study is to evaluate the safety and the maximum-tolerated dose (MTD) of the combination R-ESHAP with lenalidomide as salvage therapy for patients with relapsed or refractory diffuse large B-cell lymphoma The purpose of the Phase II of the study is to evaluate ORR of LR-ESHAP in patients with relapsed or refractory DLBCL candidates to HDT and ASCT

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL) is the most frequent subtype of non-Hodgkin's lymphoma (NHL), comprising approximately 30% of new cases. Treatment results of DLBCL have significantly improved after the introduction of rituximab (R) into CHOP-like, anthracycline-based, treatment schedules, and it is now the standard of care. Nevertheless, even with current R-CHOP-like treatment, approximately 30-40% of patients will ultimately relapse or progress.

To date, high-dose therapy (HDT) followed by autologous stem-cell transplantation (ASCT) is the reference treatment for patients with relapsed or primary refractory aggressive B-cell NHL, provided the disease is sensitive to second-line chemotherapy. Among patients with chemosensitive disease, the remission status at transplant has a significant impact on the outcome, because patients in complete remission (CR) before HDT achieve better long-term progression-free survival (PFS) than patients who undergo transplantation in partial remission (PR). Standard salvage chemotherapy for aggressive lymphoma does not exist. Commonly used second-line regimens include dexamethasone, cytarabine, cisplatin (DHAP), ESHAP (etoposide, methylprednisone, cytarabine, cisplatin), mini-BEAM (carmustine, etoposide, cytarabine, melphalan) and ICE (ifosfamide, carboplatin, etoposide). These regimens produce an overall response rate (ORR) of around 60%, and CR rates of 25% to 35%. More effective salvage regimens are needed in order to maximize the number of patients in CR prior to ASCT.

Increasing evidence suggests that rituximab added to salvage chemotherapy improves response rates and outcomes in relapsed DLBCL. In a recent randomized phase 3 study, the efficacy of adding rituximab to the DHAP-VIM-DHAP regimen was tested in 239 rituximab-naïve patients with relapsed or primary refractory aggressive cluster of differentiation 20 (CD20)+ B-cell NHL. In 225 evaluable patients, the addition of rituximab to second-line chemotherapy resulted in a significant improvement of ORR (75% versus 54%, p=.01) and PFS (52% versus 31% at two years, p<.002). Other small phase II trials (with a range of 35-55 patients) investigating rituximab in combination with ICE, DHAP or EPOCH have also shown encouraging results. However, the patients in these studies had not been previously exposed to rituximab, while at present, almost all patients with aggressive B-cell NHL receive rituximab combined with first-line chemotherapy.

In a recent multicenter retrospective study, we analyzed the influence of prior exposure to rituximab on response rates and outcomes in 163 patients with relapsed or refractory DLBCL who received Rituximab-ESHAP (R-ESHAP) as salvage therapy with a curative purpose. In this study, prior exposure to rituximab did not have an independent effect on response rates to R-ESHAP. However, a high proportion (57.4%) of patients who had received prior rituximab treatment experienced disease relapse or progression, that translated into a significantly worse PFS (17 v 57% at 3 years) and OS (38% v 67% at 3 years) as compared with rituximab-naïve patients. This observation was independent of other prognostic factors with an impact upon these outcomes, such as disease status at R-ESHAP, age-adjusted International Prognostic Index (IPI) or response to R-ESHAP. Results of the CORAL randomised trial comparing R-ICE with R-DHAP in 396 patients with relapsed or refractory DLBCL confirmed that exposure to rituximab prior to salvage therapy is associated with a worse outcome . Rituximab naïve patients had a 83% response rate and 47% 3-year event-free survival (EFS) compared with a 51% response rate and 21% EFS for patients who had received prior rituximab treatment.

These results suggest that the use of highly effective rituximab-containing primary therapy in DLBCL makes it more difficult to salvage patients who are refractory or who relapse. Thus, prospective studies incorporating new agents are needed for these patients.

Lenalidomide:

Lenalidomide, an analog of thalidomide, is a promising new therapeutic agent that does not seem to cause significant somnolence, constipation, and neuropathy, which are usually dose-limiting for thalidomide. It has been hypothesized that the mechanism of action of lenalidomide includes immunomodulatory, antineoplastic, anti-angiogenic and pro-erythropoietic properties. Preclinical as well as clinical observations demonstrate that lenalidomide downregulates production of various critical prosurvival cytokines in the tumour microenvironment while concurrently promoting activation of T- and natural killer (NK) cell-mediated antitumour response. In aggressive lymphomas, lenalidomide was shown to exert antiproliferative activity by enhancing the expression of cell cycle regulators, including p21 and SPARC, to induce G1 cell cycle arrest, caspase activation, and apoptosis.

In a recent phase II multicenter trial, 49 patients with relapsed or refractory aggressive NHL (diffuse large B-cell, follicular center grade 3, mantle cell, and transformed lymphomas) received oral lenalidomide monotherapy, 25 mg once daily on days 1 to 21, every 28 days, for 52 weeks, until disease progression or intolerance. The most common histology was diffuse large B-cell lymphoma. The median age was 65 years (range: 23 to 86). Patients had received a median of four prior treatment regimens; 56% were refractory to last therapy and 29% had received a prior ASCT. An objective response rate of 35% was observed in 49 treated patients, including a 12% rate of complete response/unconfirmed complete response. Responses were observed in each aggressive histologic subtype tested (19% ORR in patients with DLBCL). Of patients with stable disease or partial response at first assessment, 25% improved with continued treatment. Estimated median duration of response was 6.2 months, and median PFS was 4.0 months. The most common grade 4 adverse events were neutropenia (8.2%) and thrombocytopenia (8.2%); the most common grade 3 adverse events were neutropenia (24.5%), leukopenia (14.3%), and thrombocytopenia (12.2%). The results of this study show that lenalidomide monotherapy is active in relapsed or refractory aggressive NHL, with manageable side effects.

A confirmatory international phase II trial (NHL-003) of single-agent lenalidomide was performed for patients with relapsed/refractory aggressive NHL that had received at least one prior treatment and had measurable disease. Patients received 25 mg oral lenalidomide once daily on days 1-21 of every 28-day cycle and continued therapy until disease progression or toxicity. 217 patients enrolled and received lenalidomide. The ORR was 35% (77/217), with 13% (29/217) CR, 22% (48/217) PR, and 21% (45/217) with stable disease. The ORR for DLBCL was 28% (30/108), 42% (24/57) for mantel-cell lymphoma, 42% (8/19) for grade 3 follicular lymphoma, and 45% (15/33) for peripheral T-cell lymphoma. Median progression-free survival for all 217 patients was 3.7 months [95% confidence interval (CI) 2.7-5.1]. For 77 responders, the median response duration lasted 10.6 months (95% CI 7.0-NR). Median response duration was not reached in 29 patients who achieved a CR and in responding patients with follicular lymphoma (FL)-III or mantle cell lymphoma (MCL). The most common adverse event was myelosuppression with grade 4 neutropenia and thrombocytopenia in 17% and 6%, respectively.The results of this international study confirm that lenalidomide is active in heavily pre-treated patients with relapsed or refractory DLBCL with manageable side effects.

The results from these phase II studies demonstrate the activity of oral lenalidomide monotherapy in patients with relapsed or refractory aggressive NHL and warrant further investigation of lenalidomide therapy, alone or in combination, in the treatment of patients with aggressive NHL. It was recently reported that when used in combination, lenalidomide (maximum-tolerated dose [MTD] 20 mg/day, 21 of 28 days) and rituximab produce a robust response rate in relapsed or refractory mantle cell lymphoma, with a favourable toxicity profile. In multiple myeloma (MM) patients, several phase 1/2 trials have evaluated lenalidomide in conjunction with chemotherapy, such as melphalan and prednisone (MTD 10 mg/day, 21 days every 4 to 6 weeks), doxorubicin and dexamethasone (MTD 25 mg/day with G-Colony-stimulating factors (CSF), 21 of 28 days), or doxorubicin, vincristine and dexamethasone (MTD 10 mg/day, 21 days every 4 to 6 weeks). These combinations provide a considerable proportion of high-quality responses with substantial durability in patients with MM and overcomes several well-known adverse prognostic factors. A phase 1 study showed that lenalidomide can be safely combined with R-CHOP (R2CHOP) in the initial chemotherapy for aggressive B-cell lymphomas. Preliminary results of ongoing phase 2 suggest that the addition of lenalidomide to rituximab, cyclophosphamide, adriamycin, vincristine and prednisone (RCHOP) could overcome the negative prognostic impact of the non-germinal center B-cell (GCB) phenotype on outcome.

Thus, we propose an open-label, non-randomized, multicentre, escalating-dose, Phase I trial, to investigate the safety and the maximum-tolerated dose of the combination R-ESHAP with lenalidomide as salvage therapy for patients with relapsed or refractory diffuse large B-cell lymphoma candidates to stem-cell transplantation. We expect haematological toxicity as the main form of toxicity, as shown in previous studies. We must also take into account the possible adverse influence of lenalidomide treatment on stem cell mobilization. In patients with MM, prior lenalidomide therapy has been associated with high rates of failure in stem cell mobilization with filgrastim. Remobilization with chemotherapy and filgrastim is usually successful in these patients.

After selection of the maximum-tolerated dose of the combination R-ESHAP with lenalidomide a phase 2 of the study will be performed in order to evaluate the ORR of LR-ESHAP.

Partial data verification will be performed. A Clinical Research Organization (Dynamic Science S.L) Standard Operating Procedures will be used to manage the clinical trial.

Categorical variables were show by absolute and relative frequencies, including the confidence interval of 95%.

For the description of the continuous variables will be use the mean, standard deviation, median, mode, minimum and maximum, including the total number of valid values.

In the case of compare subgroups of patients, will be use for quantitative variables parametric tests or nonparametric as characteristics of the variables under study. For qualitative variables will be use Chi-square test.

Statistical analysis was planned with the Statistical Analysis System (SAS) package version 9.1 or later.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must, at the investigator's opinion, be able to meet all requirements of the clinical trial.
2. Patients must give voluntarily informed consent before performing any test test that is not part of routine care of patients.
3. Age between 18 and 70 years.
4. Candidate for treatment with high-dose QT and HSCT .
5. Diffuse large B-cell lymphoma (LDCGB) histological diagnosis according to the WHO classification ( see Annex 8).
6. Refractory lymphoma or relapsed after 1st line treatment consisting of rituximab combined with a regimen of chemotherapy (CT scan ) including anthracyclines. :

   Relapse is defined as recurrence of lymphoma after obtaining complete response (RC) with 1st line treatment . In these cases, LDCGB histologic confirmation at the time of relapse is recommended

   Refractory lymphoma be considered if it meets one of the following criteria :

   partial response after at least 6 cycles of 1st line regimen . They may also include patients in partial response after 4 cycles if the researcher believes that the response is suboptimal, and patients with stage I- II if they have received 3 cycles of R- QT + affection field radiotherapy .

   stable disease after at least 3 cycles of 1st line regimen . progression during treatment of 1st line , defined as response criteria for malignant lymphoma 2007 (see Annex 9)
7. CT scan evidence of at least two clearly demarcated lesions with a diameter of 1.5 cm, or 1 well-defined lesion with a diameter > 2 cm .
8. Evidence of positive lesions by PET, coincident with the anatomical areas affected by CT scan .
9. Eastern cooperative oncology group performance status (ECOG) less than or equal to 2.
10. Resolution of toxicities caused by the 1st line regimen to less than or equal to grade 1.
11. Women of childbearing age ( see Appendix 12) must: Obtain a negative pregnancy test before starting medically supervised therapy study. Must accept continuing pregnancy tests conducted during the course of the study and after the end of study therapy . This applies even if the patient practices complete and continued abstinence .

They must either commit to continued abstinence or heterosexual sex (which should be reviewed monthly ) or agree to use and be capable of complying with effective contraception without interruption, 28 days before starting the study drug during the study therapy (including during periods of dose interruptions ) , and for 28 days after discontinuation of study therapy .

12 male patients ( see Appendix 12) must:

* Accept to use a latex condom during any sexual relations with women of childbearing potential , even if they have had a vasectomy , while participating in this study, during dose interruptions and after discontinuation of treatment .
* Accept refrain from donating sperm while participating in this study and for a time after cessation of treatment (see specific data ) . 13. All patients must: Understand that the study drug could potentially have a teratogenic risk . Agree to abstain from donating blood while they are taking the treatment and after discontinuation of study drug therapy .

Agree not to share study medication with anyone else. For advice on precautions against pregnancy and potential risks of fetal exposure

Exclusion Criteria:

1. Patients that previously received any antitumor agent for the treatment of LDCGB except : I ) rituximab in combination with regimen including anthracyclines II ) radiotherapy as part of first-line treatment .

2 Previously received any of the following treatments in the 28 days prior to the test regime : I ) antitumor chemotherapeutic agents ; II ) radiotherapy , unless limited to a maximum dose of < or =10 Gy to control severe life-threatening symptoms ; III ) glucocorticoid except equivalent doses < or = 1 mg / kg of prednisolone / day with duration < or = 7 days; iv ) any therapeutic agent under investigation.

3. Known involvement of the central nervous system (CNS) by lymphoma. 4. Presence of abnormal or clinically significant cardiac disease, such as acute myocardial infarction or unstable angina within 6 months prior to initiation of treatment with LR- ESHAP , grade III or IV heart failure, uncontrolled hypertension or history of poor compliance with antihypertensive treatment , uncontrolled treated arrhythmias, except , with the exception of extra systoles or minor conduction abnormalities.

5. Any other serious or uncontrolled medical condition , such as diabetes, uncontrolled active infection, significant cerebrovascular disease, poorly controlled psychiatric disease, etc. .

6. Known or suspected hypersensitivity to any of the agents of the treatment under evaluation.

7. Presence of any limitations that compromise the patient's ability to comply with treatment .

8. Positive serology for HIV or Hepatitis B Virus (HBV) surface antigen (HBsAg ) . If negative for HBsAg but HBcAb positive and HBsAb negative, a HB DNA test will be performed and if positive the subject will be excluded. Note: If HBcAb positive and HBsAb positive, which is indicative of a past infection, the subject can be included 9. Active Hepatitis C (RNA positive serum) . If RNA positive result would exclude the patient from the trial in cases of patients with positive serology for Hepatitis C Virus (HCV). If the load ( RNA ) were HCV negative patients could be included in the study.

10. Prior history of malignancy other than to LDCGB (except basal or squamous cell skin and in situ carcinoma of the cervix or breast ) unless the patient free of disease beyond 5 years are.

11 Changes in laboratory values ??that might involve unacceptable risks or compromise compliance with the protocol , including: platelets < 50 x 109 / L or neutrophils <1 x 109 / L , unless attributed to infiltration by lymphoma bone marrow (MO) .

or creatinine > 1.5 times the normal upper limit . or Total bilirubin > 2 times the upper limit of normal or alanine aminotransferase (ALT) > 2.5 times the normal upper limit or alkaline phosphatase > 2.5 times the normal upper limit , unless it is attributed to hepatic infiltration by lymphoma.

12. Pregnant or breast-feeding. 13. Females of childbearing potential who do not agree to undergo pregnancy tests or repeated use effective birth control while included in the clinical trial.

14. Males patients (whose sexual partners are women of childbearing potential ) that not accept use effective birth control methods while included in the clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Phase I of the study: to evaluate the safety and the maximum-tolerated dose (MTD) of the combination R-ESHAP with lenalidomide as salvage therapy for patients with relapsed or refractory diffuse large B-cell lymphoma (determine maximum tolerated dose) | During 3 cycles of treatment (2 months after the initiation of study treatment)
  To determine the MTD of the combination R-ESHAP with lenalidomide
Phase II of the study: Phase II: to evaluate ORR of LR-ESHAP in patients with relapsed or refractory DLBCL candidates to HDT and ASCT (determine the overall response rate) | After 3 cycles of treatment (2 months after the initiation of study treatment)
  To determine the overall response rate of LR-ESHAP

SECONDARY OUTCOMES:
Phase I of the study: to analyze the adverse events of LR-ESHAP (frequency and severity of the adverse events) | During study treatment period (3 cycles of LR-ESHAP and ASCT) until end of treatment visit (3 months after ASCT)
  To describe the frequency and severity of the adverse events observed with LR-ESHAP regimen
Phase I of the study: preliminarily analyze effectiveness (response rates (CR and PR), duration of response and survival (DFS and OS) | After 3 cycles of treatment (two months after the initiation of the study treatment) and during follow-up period (36 months)
  To determine response rates (CR and PR), duration of response and survival (DFS and OS)
Phase I of the study: evaluate haematopoietic progenitor cells mobilization after treatment with LR-ESHAP (Evaluate CD34+ cell count) | After cycle 2 (5 weeks after the initiation of study treatment) or cycle 3 (9 weeks after the initiation of study treatment)
  Evaluate CD34+ cell count after treatment with LR-ESHAP
Phase I of the study: evaluate hematologic recovery after HSCT (recovery of blood parameters) | After HSCT (between 5 and 8 weeks after the initiation of the cycle 3 of treatment)
  To evaluate the recovery of blood parameters after HSCT
Phase II of the study: analyze effectiveness (Complete remission (CR) rate (determined by positron emission tomography [PET]/CT), event-free survival (EFS) and overall survival (OS) | After 3 cycles of treatment (2 months after the initiation of the study treatment) and during follo-up period (36 months)
  Complete remission (CR) rate (determined by positron emission tomography [PET]/CT), event-free survival (EFS) and overall survival (OS).
Phase II of the study: rate of transplanted patients (number of patients that undergo HSCT) | 6-8 weeks aftter the initiation of cycle 3
  To determine the number of patients that undergo HSCT
Phase II of the study: to analyze the adverse events of LR-ESHAP and ASCT. (frequency and severity of the adverse events) | During study treatment period (3 cycles of LR-ESHAP and ASCT) until end of treatment visit (3 months after ASCT)
  To describe the frequency and severity of the adverse events observed with LR-ESHAP regimen and ASCT
Phase II of the study: evaluate mobilization after treatment with LR-ESHAP (number of stem cells (2 x 106/Kg Hematopoietic progenitor cell antigen (CD34)+ cells) collected after the salvage therapy.) | After cycle 2 (5 weeks after the initiation of study treatment) or cycle 3 (9 weeks after the initiation of study treatment)
  number of stem cells (2 x 106/Kg CD34+ cells) collected after the salvage therapy.
Phase II of the study: influence of clinical and biological prognostic factors on response rates and survival (influence of clinical and biological (such as cell of origin) prognostic factors on response rates and survival.) | During study treatment (2 months) until end of treatment visit (3 months after ASCT) and during follow-up period (36 months)
  Influence of clinical and biological (such as cell of origin) prognostic factors on response rates and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Martin, Principal Investigator — University of Salamanca; Dolores Caballero, Principal Investigator — University of Salamanca
Locations (9):
- Spain (9):
  - ICO- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - ICO- Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Alejandro Martín, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario La Fe, Valencia

REFERENCES:
- [Background] Harting R, Venugopal P, Gregory SA, O'brien T, Bogdanova E. Efficacy and safety of rituximab combined with ESHAP chemotherapy for the treatment of relapsed/refractory aggressive B-cell non-Hodgkin lymphoma. Clin Lymphoma Myeloma. 2007 May;7(6):406-12. doi: 10.3816/CLM.2007.n.019. PMID 17621406
- [Background] Feldman T, Mato AR, Chow KF, Protomastro EA, Yannotti KM, Bhattacharyya P, Yang X, Donato ML, Rowley SD, Carini C, Valentinetti M, Smith J, Gadaleta G, Bejot C, Stives S, Timberg M, Kdiry S, Pecora AL, Beaven AW, Goy A. Addition of lenalidomide to rituximab, ifosfamide, carboplatin, etoposide (RICER) in first-relapse/primary refractory diffuse large B-cell lymphoma. Br J Haematol. 2014 Jul;166(1):77-83. doi: 10.1111/bjh.12846. Epub 2014 Mar 25. PMID 24661044
- [Background] Chiappella A, Tucci A, Castellino A, Pavone V, Baldi I, Carella AM, Orsucci L, Zanni M, Salvi F, Liberati AM, Gaidano G, Bottelli C, Rossini B, Perticone S, De Masi P, Ladetto M, Ciccone G, Palumbo A, Rossi G, Vitolo U; Fondazione Italiana Linfomi. Lenalidomide plus cyclophosphamide, doxorubicin, vincristine, prednisone and rituximab is safe and effective in untreated, elderly patients with diffuse large B-cell lymphoma: a phase I study by the Fondazione Italiana Linfomi. Haematologica. 2013 Nov;98(11):1732-8. doi: 10.3324/haematol.2013.085134. Epub 2013 Jun 28. PMID 23812930
- [Background] Nowakowski GS, LaPlant B, Habermann TM, Rivera CE, Macon WR, Inwards DJ, Micallef IN, Johnston PB, Porrata LF, Ansell SM, Klebig RR, Reeder CB, Witzig TE. Lenalidomide can be safely combined with R-CHOP (R2CHOP) in the initial chemotherapy for aggressive B-cell lymphomas: phase I study. Leukemia. 2011 Dec;25(12):1877-81. doi: 10.1038/leu.2011.165. Epub 2011 Jul 1. PMID 21720383
- [Background] Wang M, Fowler N, Wagner-Bartak N, Feng L, Romaguera J, Neelapu SS, Hagemeister F, Fanale M, Oki Y, Pro B, Shah J, Thomas S, Younes A, Hosing C, Zhang L, Newberry KJ, Desai M, Cheng N, Badillo M, Bejarano M, Chen Y, Young KH, Champlin R, Kwak L, Fayad L. Oral lenalidomide with rituximab in relapsed or refractory diffuse large cell, follicular and transformed lymphoma: a phase II clinical trial. Leukemia. 2013 Sep;27(9):1902-9. doi: 10.1038/leu.2013.95. Epub 2013 Apr 2. PMID 23545991
- [Derived] Martin Garcia-Sancho A, Baile M, Rodriguez G, Dlouhy I, Sancho JM, Jarque I, Gonzalez-Barca E, Salar A, Espeso M, Grande C, Bergua J, Montes-Moreno S, Redondo A, Enjuanes A, Campo E, Lopez-Guillermo A, Caballero D. Lenalidomide in combination with R-ESHAP in patients with relapsed or refractory diffuse large B-cell lymphoma: A phase 2 study from GELTAMO. Br J Haematol. 2023 Oct;203(2):202-211. doi: 10.1111/bjh.18989. Epub 2023 Jul 23. PMID 37485564
- See also: Sponsor web page — http://www.geltamo.com/